CLINICAL TRIAL: NCT07326670
Title: Comparison of Spinal and General Anesthesia on Systemic Inflammatory Response in Patients Undergoing Percutaneous Nephrolithotomy: Evaluation of SII, SIRI, AISI, NLR, and RDW
Brief Title: Effects of Spinal vs General Anesthesia on Systemic Inflammation in PCNL
Acronym: PCNL-ANES-INF
Status: Recruiting | Type: Observational
Sponsor: Elazıg Fethi Sekin Sehir Hastanesi (Other)
Responsible Party: Principal Investigator, Sevim Şenol Karataş, Specialist in Anesthesiology and Reanimation, Elazıg Fethi Sekin Sehir Hastanesi
Other Study IDs: PCNL-ANES-INFLAM-2025
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Anesthesia Techniques; Percutaneous Nephrolithotomy; Systemic Inflammation
Keywords: Percutaneous nephrolithotomy; Spinal anesthesia; Neutrophil-to-lymphocyte ratio; Red cell distribution width; Systemic inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spinal Anesthesia Group: Patients undergoing percutaneous nephrolithotomy under spinal anesthesia as part of routine clinical practice. No additional intervention is performed for the purposes of the study.
- General Anesthesia Group: Patients undergoing percutaneous nephrolithotomy under general anesthesia as part of routine clinical practice. No additional intervention is performed for the purposes of the study.

SUMMARY:
This observational study aims to compare the effects of spinal and general anesthesia on perioperative systemic inflammatory response in patients undergoing percutaneous nephrolithotomy (PCNL). Systemic inflammatory indices derived from routine complete blood count parameters, including Systemic Immune-Inflammation Index (SII), Systemic Inflammation Response Index (SIRI), Aggregate Index of Systemic Inflammation (AISI), Neutrophil-to-Lymphocyte Ratio (NLR), and Red Cell Distribution Width (RDW), will be evaluated. Preoperative and postoperative laboratory values will be analyzed to determine whether the type of anesthesia influences systemic inflammatory markers and related clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status class I-III
* Patients aged 18 years and older

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status class IV or V
* Patients younger than 18 years
* Active infection or diagnosis of sepsis
* Malignancy
* Chronic inflammatory diseases (e.g., rheumatoid arthritis, systemic lupus erythematosus)
* Use of immunosuppressive therapy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years and older who undergo elective percutaneous nephrolithotomy (PCNL) surgery and meet the eligibility criteria. Patients classified as American Society of Anesthesiologists (ASA) physical status I-III are included. All participants receive either spinal or general anesthesia as part of routine clinical practice, and no additional intervention is performed for research purposes.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Perioperative change in systemic inflammatory indices (SII, SIRI, AISI, NLR, RDW) | From preoperative period (within 6 hours before surgery) to postoperative period (6-24 hours after surgery)
  Changes in Systemic Immune-Inflammation Index (SII), Systemic Inflammation Response Index (SIRI), Aggregate Index of Systemic Inflammation (AISI), Neutrophil-to-Lymphocyte Ratio (NLR), and Red Cell Distribution Width (RDW) will be evaluated using routine complete blood count parameters obtained preoperatively and postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Fethi Sekin City Hospital, Elâzığ, Elaziğ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No